CLINICAL TRIAL: NCT01232062
Title: Study of High-dose Chemotherapy Combined With Adoptive Cellular Therapy With Dentritic and Cytokine-induced Killer Cells in Triple Negative Breast Cancer Patients
Brief Title: Study of High-dose Chemotherapy (HDC) Combined With Adoptive Cellular Therapy With DC-CIK Cells in Triple Negative Breast Cancer Patients
Acronym: DC-CIK
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Ren, Director, Peking University Cancer Hospital & Institute
Other Study IDs: HD+DC-CIK
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: breast neoplasm; Neoplasm Metastasis; Drug Therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — about 4ml peripheral vein blood，paraffin section on metastatic tissue，
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To access the effectiveness of High-dose Cyclophosphamide Combined Chemotherapy combined with adoptive cellular therapy with dentritic and cytokine-induced killer cells in triple negative metastatic breast cancer patients

DETAILED DESCRIPTION:
1. Metastatic breast cancer patients should be definitively diagnosis based on histopathology, with ER-negative and PR-negative, FISH testing for her-2-negative
2. All the patients enrolled will be given standard HDC and cellular therapy.HDC and cellular therapy consisting of one cycle of HDC followed by an apheresis and ex vivo cultures to generate DC and CIK. DC-CIK infusions were given to each patient, followed by two cycles HDC, plus low-dose Oral Cyclophosphamide.
3. PET-CT scans were done on each patients at baseline and after chemotherapy. The response is assessed using Response Evaluation Criteria in Solid Tumor Group (RECIST) guidelines.
4. Estimate time to progression, survival rates and clinical benefit response on patients.
5. Find biomarkers associated with drug response.

ELIGIBILITY:
Inclusion Criteria:

* Failure to anthracycline and/or taxol chemotherapy;
* metastatic tumor is histologically confirmed by immunohistochemical staining to be ER-negative and PR-negative. FISH testing for her-2-negative;
* Metastatic tumor can not be removed through surgery procedure;
* Metastatic tumor measured by PET-CT scan is at least 1cm;
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Normal cardiac, hepatic, renal and bone marrow functions;
* Life expectancy ≥3 months.

Exclusion Criteria:

* Do not finish twice PET-CT scan;
* Central nervous system metastases;
* Serious or uncontrolled concurrent medical illness;
* History of other malignancies;
* Having been enrolled in some other clinal trials within a month;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female patients with metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
response to chemotherapy | 4months
  Response to chemotherapy is evaluated by Response Evaluation Criteria in Solid Tumors(RESIST).

SECONDARY OUTCOMES:
Time to disease progression | six months to one year
  Time to disease progression is measured from the date therapy is initiated to the date of documented disease progression.
survival rates | one-year
clinical benefit response | six months to one year
  clinical benefit response include CR,PR,SD

CONTACTS AND LOCATIONS:
Overall Officials: JING YU, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; CHAO YING WANG, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; JUN REN, MD, PhD, Study Chair — Peking University Cancer Hospital & Institute; YU LIN ZHU, MD, PhD, Principal Investigator — Bei jing Cancer Hospital; Jie Zhang, MD., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China